CLINICAL TRIAL: NCT03538522
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, and Efficacy of NA-831 in Alzheimer Patients With Mild Cognitive Impairment
Brief Title: A Double-Blind, Placebo-Controlled Safety and Efficacy Study of NA-831
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomed Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NeuroActiva
Record Dates: First submitted 2018-03-16; First posted 2018-05-29 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2019-11

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Alzheimer Dementia; Dementia, Vascular; Dementia With Lewy Bodies; Cognitive Impairment; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Cognitive Disorder
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low-dose N-831(Traneurocin)- 10 mg QD (Experimental): Oral administration of 10 mg of NA-831 (Traneurocin) per day for 24 weeks
  Interventions: Drug: N-831(Traneurocin) 10 mg QD
- Medium-dose NA-831(Traneurocin)- 20 mg QD (Experimental): Oral administration of 20 mg of NA-831(Traneurocin) per day for 24 weeks
  Interventions: Drug: NA-831 (Traneurocin) 20 mg QD
- High-dose NA-831(Traneurocin)- 40 mg QD (Experimental): Oral administration of 40 mg of NA-831(Traneurocin) per day for 24 weeks
  Interventions: Drug: NA-831 (Traneurocin) 40 mg QD
- Placebo (Placebo Comparator): Oral administration of placebo per day for 24 weeks
  Interventions: Drug: Placebo oral capsule QD

INTERVENTIONS:
Drug: N-831(Traneurocin) 10 mg QD — Oral administration of 10 mg capsule of NA-831 QD for 24 weeks
  Arms: Low-dose N-831(Traneurocin)- 10 mg QD
Drug: NA-831 (Traneurocin) 20 mg QD — Oral administration of 20 mg capsule of NA-831 QD for 24 weeks
  Arms: Medium-dose NA-831(Traneurocin)- 20 mg QD
Drug: NA-831 (Traneurocin) 40 mg QD — Oral administration of 40 mg capsule of NA-831 QD or for 24 weeks
  Arms: High-dose NA-831(Traneurocin)- 40 mg QD
Drug: Placebo oral capsule QD — Oral administration of oral placebo capsule QD or 24 weeks
  Arms: Placebo

SUMMARY:
This study seeks to evaluate the efficacy and safety of NA-83 in subjects with mild cognitive impairment due to Alzheimer's Disease

DETAILED DESCRIPTION:
Mild cognitive impairment ("MCI") is defined as the "symptomatic pre-dementia stage" on the continuum of cognitive decline. Currently, no medications have proven effective for MCI. Preclinical experiments indicate that NA-831 is an endogenous small molecule that exhibits neuroprotection, neurogenesis, and cognitive protective properties across a range of disease models. NA-831 has been shown to be safe and well tolerated in healthy volunteers. This study seeks to evaluate the efficacy and safety of NA-83 in 126 subjects with mild cognitive impairment due to Alzheimer's Disease

ELIGIBILITY:
INCLUSION

1. Is male or female, at 55-85 years of age (inclusive) at screening self-reported memory complaint, corroborated by spouse or companion as appropriate.
2. Wechsler Memory Scale III (WMS-III) age-adjusted Logical Memory II score ≤ 5.
3. Mini-Mental State Exam (MMSE) ≥23
4. Center for Epidemiologic Studies-Depression (CES-D) score <27.
5. Normal thyroid function, defined as TSH, T3 and T4 within normal limits.
6. Agree not to consume alcoholic beverages within 8 hours of each study visit.
7. Willing and able to sign informed consent and complete the CTB and all other tests and procedures as listed in the protocol.
8. Able to read at a 6th grade level or equivalent
9. Female subjects must be surgically sterile or post-menopausal for at least 2 years. If <2 years post-menopausal, then a follicle stimulating hormone (FSH) ≥40 mIU/mL must be obtained.
10. If participant is receiving an acetylcholinesterase inhibitor or memantine, the dose must have been stable for at least three months before Screening
11. Must have a reliable and competent trial partner/informant who has a close relationship with the participant and is willing to accompany the participant to all required trial visits, and to monitor compliance of the administration of the trial medication

EXCLUSION CRITERIA

1. Subjects who have any significant, untreated psychiatric illness or any CNS condition (such as schizophrenia, Parkinson's disease, stroke, etc.) that could interfere with the study evaluations or procedures or which poses an additional risk.
2. Evidence of a clinically relevant or unstable psychiatric disorder, excluding major depression in remission
3. History of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.
4. Have had a stroke or Transient Ischemic Attack (TIA) or unexplained loss of consciousness in the past 1 year
5. History of seizures or epilepsy within the last 5 years
6. History of hepatitis or liver disease that has been active within the 6 months prior toScreening
7. History of malignancy occurring within the 5 years before Screening, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or localized prostate carcinoma
8. Clinically significant vitamin B12 or folate deficiency in the 6 months before Screening
9. History of unstable angina, myocardial infarction, chronic heart failure or clinically significant conduction abnormalities within 1 year prior to Screening Visit
10. History of alcohol or substance abuse or dependence within the past year.
11. Has human immunodeficiency virus (HIV) by medical history
12. Acute infective sinusitis.
13. History or presence of an abnormality of the external or internal structures of the nose or nasopharynx, except for surgical correction of the nasal septum or a "broken nose" at least 2 years previously, or surgical repair of cleft palate when <30 years of age.
14. Use of medications that are known to cause frank obtundation of cognition
15. History of or current significant systemic disease judged to interfere with the study evaluations or likely to be a safety concern.
16. Untreated sleep apnea or treatment for sleep apnea for <3 months.
17. Clinically significant systemic illness or serious infection within 30 days prior to or during the screening period
18. Use of allowed medications for chronic conditions at doses that have not been stable for at least 4 weeks prior to Screening, or use of AD medications at doses that have not been stable for at least 8 weeks prior to Screening
19. Abnormal clinical laboratory test results, specifically: Alanine transaminase (ALT) or aspartate transaminase (AST) >2 х the upper limit of normal (ULN),Hematology <80% the lower limit of normal, Creatinine ≥2 mg/dL and ,Other clinical laboratory values or vital signs considered clinically significant in the opinion of the Investigator.
20. Treatment with any investigational drug, biologic, or device within the previous 30 days prior to screening.
21. Surgery involving general anesthesia within the past 3 months or planned surgery requiring general anesthesia during the study period.
22. Contraindications to study procedures
23. Use of any medications that, in the opinion of the Investigator, may contribute to cognitive impairment, put the participants at higher risk for adverse events (AEs), or impair the participant's ability to perform cognitive testing or complete study procedures.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Clinical Dementia Rating Scale- Sum of Boxes (CDR-SB) score at Week 24 | Week 24
  To study to the change from baseline in the Clinical Dementia Rating scale-Sum of Boxes (CDR-SB) score at Week 2 and Week 24.
  The CDR-SB is obtained through interviews of patients and informants, and cognitive functioning is rated in 6 domains of functioning: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a 5-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). The CDR-SOB score is obtained by summing each of the domain box scores, with scores ranging from 0 to 18 with the higher values represent worse outcome.

SECONDARY OUTCOMES:
1. Mean difference between the last (Week 24) and first (Week 2) postdose using Clinical Dementia Rating Scale- Sum of Boxes (CDR-SB) assessment | Week 24
  To assess the Clinical Dementia Rating Scale- Sum of Boxes (CDR-SB) mean difference between the Week 2 and Week 24.
  The CDR-SB is obtained through interviews of patients and informants, and cognitive functioning is rated in 6 domains of functioning: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a 5-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). The CDR-SOB score is obtained by summing each of the domain box scores, with scores ranging from 0 to 18, with the higher values represent worse outcome.
Assess the change from baseline in ADCS-ADL MCI at Week 24 | Week 24
  Change from baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (Mild Cognitive Impairment version) (ADCS-ADL MCI) at Week 24.
  The Galasko method for Alzheimer Disease Cooperative Study (ADCS) will be used, which contains 23 items covering physical and mental functioning and independence in self-care. For Activities of Daily Living (ADLs), the scoring used was the following: 0 = no impairment, 1 = problem performing but no supervision or assistance needed, 2 = problem requiring supervision, 3 = problem with assistance needed, and 4 = unable to perform.
  The scores range from 0 to 78, with higher values indicates greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd Tran, PhD, Study Director — Biomed Industries, Inc.
Locations (2):
- New Zealand (2):
  - NeuroActiva-Clinical Research Unit, Auckland
  - NeuroActiva Testing Facility of NeuroActiva (New Zealand) Ltd, Auckland

IPD SHARING:
Plan to Share IPD: Undecided